CLINICAL TRIAL: NCT00274183
Title: Prevalence, Clinicopathological Characteristics, Biomarkers and Genetics of Nonalcoholic Steatohepatitis in Taiwanese Children
Brief Title: Nonalcoholic Fatty Liver Disease in Taiwanese Children
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 94034
Record Dates: First submitted 2006-01-02; First posted 2006-01-10 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2018-12

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, WBC DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is an emerging and important disease in Taiwan. However, the prevalence and clinical characteristics have not been studied well. The purpose of this study is to resolve the aforementioned problem.

DETAILED DESCRIPTION:
[Study Subjects] Obesity was defined as the BMI value > 95 percentile by different age- and gender groups according to the standards of the Department of Health in Taiwan.

[Data Collection] The following data were obtained for each subject: age, gender, BMI, waist and hip circumference. BMI was calculated as body weight (kg)/ height (m2).

In fasting venous blood samples, we measured total serum bilirubin, alanine aminotransferase, aspartate aminotransferase, γ-glutamyltransferase, fasting glucose, triglyceride, total cholesterol,high-density lipoprotein cholesterol, insulin, glucose, and adiponectin.

[Liver Ultrasonography] All participants underwent an ultrasonographic study of the liver performed by one operator.

NAFLD was defined as the presence of an ultrasonographic pattern consistent with the following criteria: liver-kidney echo discrepancy, attenuated echo penetration and visibility of diaphragm, and obscure hepatic vessel structures.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of fatty liver

Exclusion Criteria:

* other hepatic diseases

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Obese children will be enrolled from elementary school and high school in Taiwan
Sampling Method: Probability Sample
Enrollment: 614 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
non-alcoholic fatty liver disease | one year
  confirmed by liver ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Lin, M.D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin YC, Chang PF, Chang MH, Ni YH. Genetic variants in GCKR and PNPLA3 confer susceptibility to nonalcoholic fatty liver disease in obese individuals. Am J Clin Nutr. 2014 Apr;99(4):869-74. doi: 10.3945/ajcn.113.079749. Epub 2014 Jan 29. PMID 24477042
- [Derived] Lin YC, Chang PF, Chang MH, Ni YH. A common variant in the peroxisome proliferator-activated receptor-gamma coactivator-1alpha gene is associated with nonalcoholic fatty liver disease in obese children. Am J Clin Nutr. 2013 Feb;97(2):326-31. doi: 10.3945/ajcn.112.046417. Epub 2012 Dec 26. PMID 23269818